CLINICAL TRIAL: NCT02266849
Title: Loperamide vs. Placebo's Effect on Ileostomy Output: A Clinical Randomized Blinded Cross-over Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insuficcient recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Niels Qvist, Professor, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: s-20140081
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Rectal Cancer; Ulcerative Colitis; Short Bowel Syndrome
MeSH Terms: conditions — Rectal Neoplasms; Colitis, Ulcerative; Short Bowel Syndrome | interventions — Loperamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loperamide (Active Comparator): Patients will take the drug for three days. Day 1 - uploading with the drug Day 2 - collecting output when necessary Day 3 - radiopaque marker and collection of output every two hours
  Interventions: Drug: Loperamide
- Placebo (Placebo Comparator): Patients will take the drug for three days. Day 1 - uploading with the drug Day 2 - collecting output when necessary Day 3 - radiopaque marker and collection of output every two hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Loperamide — 12 mg Loperamide each day for three days
  Other Names: Imodium
  Arms: Loperamide
Drug: Placebo — 6 tablets daily for three days
  Arms: Placebo

SUMMARY:
Clinical experience show limited effect of the drug Loperamide used to decrease output in stoma patients. Therefore the investigators see the need for a randomized blinded clinical trial to determine the effect of Loperamide opposite Placebo.

Loperamide will be evaluated in relation to the following parameters

* Change in ileostomy output in g/day in relation to oral intake
* Quantification of the change in intestinal transit time using a radiopaque marker
* The patient´s own assessment on which period they received Loperamide or Placebo

DETAILED DESCRIPTION:
The aim of this study is to quantify the effect of Loperamide on ileostomy output in patients operated for rectal cancer, ulcerative colitis and in patients with short bowl syndrome. These patients are recruited through The Department of Surgery and The Department of Gastroenterology, University Hospital Odense. The effect of Loperamide will be evaluated against Placebo in relation to the following parameters:

* Change in ileostomy output in g/day in relation to oral intake
* Quantification of the change in intestinal transit time using a radiopaque marker
* The patient´s own assessment on which period they received Loperamide or Placebo

Construction of a stoma is a frequently used part of the surgical treatment of intestinal cancer and chronic intestinal inflammation. More than 60% of patients with an ileostomy develop dehydration and loss of salts and minerals, due to an excessive stoma output. The most common method used to reduce stoma output is Imodium® ( Loperamide ). The effect has never been studied extensively, probably because it is an over the counter medicine. The treatment is relatively expensive and also subject to side effects, even if they are mild. Therefore, the investigators found it relevant to perform a clinical study to determine the effect. The results will be important for future patient treatment.

The study is a clinical blinded randomized crossover study. The study includes three types of patients. Patients operated for rectal cancer or ulcerative colitis with a temporary or permanent ileostomy, and patients with short bowel syndrome with a permanent ileostomy. The first two types of patients will be recruited through two ways.

* During hospitalization in connection to their operation at The Department of Surgery, University Hospital Odense. The patients are offered inclusion into the study either before or after surgery depending upon the clinical situation. For those who consent and fulfills the inclusion criteria, the study starts up on 7th day after surgery.
* Through their regular controls in the stoma clinic.

Patients with short bowel syndrome are offered inclusion through their contact with The Department of Gastroenterology, University Hospital Odense, if they meet the criteria for inclusion.

Patients will undergo to periods during the study. They will be randomized to start with either Loperamide or Placebo. Each period consists of 3 days.

Day 1 - Uploading of the drug

Day 2 - Collecting of stoma output when necessary

Day 3 - Radiopaque marker and collection of stoma output every two hours

After 7 days without medicine intake the patient starts the second period with the opposite drug.

During day 2-3 the patient will register and weigh all food and fluid intake.

ELIGIBILITY:
Inclusion Criteria:

* Operation for rectal cancer or ulcerative colitis an ileostomy (loop or end ileostomy within the last 7 days) OR
* ileostomy patient with contact to the stoma clinic OR
* Short bowel syndrome with a permanent ileostomy
* signed consent form

Exclusion Criteria:

* Complications associated with surgery
* Non-radical surgery
* Chemotherapy
* Poor compliance
* Other serious illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Output weight | 2 days
  Collection af output for two days to compare between the two periods

SECONDARY OUTCOMES:
Gastrointestinal transit time | 10 hours
  Patients swallow a pill with radiopaque markers and collect stoma output every two hours

OTHER OUTCOMES:
Patient evaluation | 14 days
  Patients evaluation on when they received Loperamide and Placebo at the end of the collecting period

CONTACTS AND LOCATIONS:
Overall Officials: Niels Qvist, MD, DMsc, Study Director — Odense University Hospital, Department of Surgery A, Denmark
Locations (1):
- Odense University Hospital, Surgical Department A, Odense, Denmark

REFERENCES:
- [Derived] Kristensen K, Qvist N. The Acute Effect of Loperamide on Ileostomy Output: A Randomized, Double-Blinded, Placebo-Controlled, Crossover Study. Basic Clin Pharmacol Toxicol. 2017 Dec;121(6):493-498. doi: 10.1111/bcpt.12830. Epub 2017 Jul 10. PMID 28627732